CLINICAL TRIAL: NCT00973804
Title: Pilot Trial of Targeted Immune-Depleting Chemotherapy and Reduced-Intensity Matched Unrelated Double Cord Blood Transplant for the Treatment of Leukemias, Lymphomas, and Pre-Malignant Blood Disorders
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090210; 09-C-0210
Record Dates: First submitted 2009-09-05; First posted 2009-09-09 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-05-20

CONDITIONS: Leukemia; Non-Hodgkins Lymphoma; Hodgkins Lymphoma; MDS; Multiple Myeloma
Keywords: Reduced Intensity Conditioning; Umbilical Cord Blood Transplant; Targeted Immune Depletion; Leukemia; Lymphoma; Multiple Myeloma; Non-Hodgkins Lymphoma; Hodgkins Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Lymphoma | interventions — Tacrolimus; Sirolimus

INTERVENTIONS:
Drug: EPOCH-F/R
Drug: FLAG
Drug: Transplant Preparative Regimen (Flu/Cy/Mes)
Drug: GVHD Prophylaxis (tacrolimus and sirolimus)
Procedure: Double Cord Blood Transplantation

SUMMARY:
Background:

* Allogeneic stem cell transplantation (SCT) has been used to treat many kinds of cancer or pre-cancerous conditions that develop in blood or immune system cells. Umbilical cord blood transplantation (UCBT) is a type of allogeneic transplant that is used when none of a patient s siblings are a match and an acceptable match cannot be identified from one of the bone marrow registries. Prior to receiving the cord blood stem cells, large doses of chemotherapy drugs and/or radiation have been traditionally used to eliminate most of the cancerous or abnormal cells from the recipient s system, along with most of his or her own stem cells and immune cells. Donor stem cells then replace the recipient s stem cells in the bone marrow, restoring normal blood production and immunity. In this way, an allogeneic SCT provides not only new blood cells but an entire new immune system.
* In the past, allogeneic SCT was performed with very high doses of chemotherapy and/or radiation to get rid of as much of the recipient s cancer as possible and prevent rejection of the treatment. However, intensive chemotherapy or radiation can cause serious side effects, including death. A newer method uses smaller, less toxic doses of chemotherapy and/or radiation before allogeneic SCT. In these reduced-intensity stem cell transplants, the recipient s stem cells and immunity are not completely eliminated, but they are weakened enough to help prevent the donor s cells from being rejected.

Objectives:

- To study the safety and effectiveness of reduced-intensity stem cell transplants given with immune-depleting chemotherapy and umbilical cord blood provided by an unrelated donor.

Eligibility:

* Individuals between 18 and 69 years of age who have been diagnosed with any of a number of cancerous and pre-cancerous blood conditions, including lymphoma and leukemia.
* Participants must not have a potential donor sibling or a readily available unrelated donor identified through one of the bone marrow donor registries.

Design:

* Patients will be matched with at least two umbilical cords with an acceptable cell dose. The two frozen umbilical cord blood units will be sent to the NIH prior to the date of transplant.
* Patients will receive one, two, or three cycles of chemotherapy (based on the type of disease) to treat the disease and to weaken the immune system. Patients who already have a weakened immune system from other treatments will not receive this round of chemotherapy.
* Patients will then receive 4 days of reduced-intensity transplant chemotherapy (also called the conditioning regimen ) to prepare for the transplant.
* Two days after transplant chemotherapy, patients will receive the transplant, with the two umbilical cords infused one after the other on the same day. Patients will receive additional treatment to prevent complications.
* Patients will remain in the hospital for 4 to 6 weeks after the transplant, and will be discharged for outpatient treatment when the study doctors deem it appropriate.
* Patients will continue on medications at home to lower the risk of complications and infections, and will visit the NIH clinic regularly for the first 6 months after the transplant, and then less often for at least 5 years afterward.

DETAILED DESCRIPTION:
Background:

The major limitations of umbilical cord blood transplantation (UCBT) in adults are graft rejection and delayed engraftment leading to increased infection-related morbidity and treatment related mortality (TRM). To increase engraftment rates while at the same time enhancing graft-versus-tumor effect, previous studies within our institution have employed the strategy of targeted immune depletion (TID). The goal of TID is to use T-cell suppressive chemotherapy prior to the conditioning regimen to treat the patient s disease while concurrently depleting host T-cells. This has lead to earlier complete donor chimerism in the setting of allogeneic sibling donor and matched unrelated donor transplantation. Our aim in the current protocol is to extend the strategy of TID to reduced-intensity UCBT, with the goal of more rapid engraftment, leading to decreased TRM and increased overall survival. Our intention is to investigate this approach in the setting of double cord blood transplant in adults in a pilot manner.

Objectives:

* The primary objective of this study is to see whether targeted immune depletion can shorten the time to neutrophil recovery and improve the cord blood engraftment rate as measured by ANC greater than or equal to 500 x 3 and at least partial donor chimerism (10-90%).
* Secondary objectives include further assessment of hematopoetic recovery, treatment related morbidity including infections and acute and chronic GVHD, TRM, progression free and overall survival, further assessment of immune reconstitution, and study of engraftment kinetics as they apply to prediction of which of the two transplanted cords will engraft in relation to cell dose, CD34+ dose, HLA-match, and other experimental variables.

Eligibility:

* Adults (18-69 years) with advanced or high-risk hematologic malignancies including AML, ALL, MDS, CLL, NHL, HL, CML, multiple myeloma, and MPD who lack a readily available HLA-matched sibling or greater than or equal to 7/8 HLA-matched unrelated donor. Patients must have life expectancy of at least 3 months, ECOG less than or equal to 2, and relatively normal major organ functions.
* Patients must have two partially HLA-matched UCB units. Units must be HLA-matched at HLA-A and B (intermediate resolution molecular typing) and DRB1 (high resolution molecular typing) 4-6/6 with the recipient and 4-6/6 with each other. Each unit must contain a minimum precryopreserved, nucleated cell dose of 1.5 x 10(7) per kilogram.

Design:

* This is a Pilot study of TID in the setting of reduced-intensity double cord blood transplant in adults.
* Patients will receive disease-specific induction chemotherapy (EPOCH-F/R or FLAG) prior to transplant for disease control and immune depletion.
* All patients will receive an identical conditioning regimen consisting of cyclophosphamide 1200 mg/m(2)/day IV for 4 days and fludarabine 30 mg/m(2)/day for 4 days.
* A maximum of 13 patients will be transplanted in the initial part of this pilot study. If no stopping rules are reached, the study will be expanded to allow the transplantation of an additional 12 patients (a total of 25 patients).

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Adults (18-69 years) with advanced or high-risk hematologic malignancies including AML, ALL, MDS, CLL, NHL, HL, CML, multiple myeloma, and MPD who lack a readily available HLA-matched sibling or greater than or equal to 7/8 HLA-matched unrelated donor. Patients must have life expectancy of at least 3 months, ECOG less than or equal to 2, and relatively normal major organ functions.
* Patients must have two partially HLA-matched UCB units. Units must be HLA-matched at HLA-A and B (intermediate resolution molecular typing) and DRB1 (high resolution molecular typing) 4-6/6 with the recipient and 4-6/6 with each other. Each unit must contain a minimum precryopreserved, nucleated cell dose of 1.5 x 10(7) per kilogram.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-08-25; Primary Completion 2013-05-20 (Actual); Study Completion 2013-05-20 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to see whether targeted immune depletion can shorten the time to hematopoietic recovery and improve cord blood engraftment rate as measured by ANC greater than 500 X 3 and at least partial donor chimerism (...

SECONDARY OUTCOMES:
Secondary objectives include further assessment of immune reconstitution, study of engraftment kinetics in relation to cell dose and HLA-match, and comprehensive assessment of acute and chronic GVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z Pavletic, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Laughlin MJ, Eapen M, Rubinstein P, Wagner JE, Zhang MJ, Champlin RE, Stevens C, Barker JN, Gale RP, Lazarus HM, Marks DI, van Rood JJ, Scaradavou A, Horowitz MM. Outcomes after transplantation of cord blood or bone marrow from unrelated donors in adults with leukemia. N Engl J Med. 2004 Nov 25;351(22):2265-75. doi: 10.1056/NEJMoa041276. PMID 15564543
- [Background] Rocha V, Labopin M, Sanz G, Arcese W, Schwerdtfeger R, Bosi A, Jacobsen N, Ruutu T, de Lima M, Finke J, Frassoni F, Gluckman E; Acute Leukemia Working Party of European Blood and Marrow Transplant Group; Eurocord-Netcord Registry. Transplants of umbilical-cord blood or bone marrow from unrelated donors in adults with acute leukemia. N Engl J Med. 2004 Nov 25;351(22):2276-85. doi: 10.1056/NEJMoa041469. PMID 15564544
- [Background] Bishop MR, Steinberg SM, Gress RE, Hardy NM, Marchigiani D, Kasten-Sportes C, Dean R, Pavletic SZ, Gea-Banacloche J, Castro K, Hakim F, Krumlauf M, Read EJ, Carter C, Leitman SF, Fowler DH. Targeted pretransplant host lymphocyte depletion prior to T-cell depleted reduced-intensity allogeneic stem cell transplantation. Br J Haematol. 2004 Sep;126(6):837-43. doi: 10.1111/j.1365-2141.2004.05133.x. PMID 15352988